CLINICAL TRIAL: NCT06805318
Title: Development and Assessment of a Vocational Rehabilitation Intervention for Job Retention in Workers With Multiple Sclerosis (RiaLSM Intervention Project)
Brief Title: Feasibility of a Vocational Rehabilitation Intervention for Job Retention in Workers With MS-RiaLSM Intervention Project
Acronym: RialSM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Italiana Sclerosi Multipla (Other)
Collaborators: Italian Multiple Sclerosis Society (AISM)Liguria, Genoa (Unknown); IRCCS Santa Lucia Foundation, Rome (Unknown); IRCCS San Martino Hospital, Genoa (Unknown); Italian Workers' Compensation Authority (INAIL) (Unknown); Department of Health Science (DiSSaL), University of Genoa, Genoa (Unknown)
Responsible Party: Principal Investigator, Michela Ponzio, PhD, Principal Investigator, Fondazione Italiana Sclerosi Multipla
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: CET Liguria:329/2024-DBid13998; Grant BRic 2022, ID 31 (Other Grant/Funding Number: Supported by INAIL - Italian Workers' Compensation Authority)
Record Dates: First submitted 2025-01-03; First posted 2025-02-03 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-01

CONDITIONS: Multiple Sclerosis; Vocational Rehabilitation
Keywords: Multiple Sclerosis; Vocational Rehabilitation; Occupational Rehabilitation; Return to Work; Work Maintenance; Work Placement; Vocational Guidance; Reasonable Accomodation
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Intervention Model Description: The study design will be an explorative interventional pilot study. Participants will be recruited in the study among workers with MS in contact with AISM (Italian Multiple Sclerosis Society) Rehabilitation Service in Liguria, and Santa Lucia Foundation IRCCS, Rome. A sample of 30 workers with job difficulties (MSQ-Job>=15) will be recruited for interventional study among subjects participating in a previous cross-sectional study.
  The VR intervention will be based on individual needs, covering three areas of intervention: the medical-rehabilitation area, the reasonable accommodation area, and the education area.
  During baseline evaluation, a maximum of 5 priority work difficulties will be identified for each subject. At the end of the VR intervention, the following aspects will be evaluated: resolution of work difficulties, satisfaction and effectiveness of the intervention through the Global Perceived Effect.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- VR intervention (Experimental): This is a single-arm study. Therefore, the intervention will be conducted on the whole sample. The nature of the rehabilitation program will vary and will cover three different areas: the rehabilitation area, the reasonable accommodation area, and the educational and formative area. Participants can receive any of the three types of intervention, or a combination of these, based on individual needs.
  Interventions: Behavioral: Vocational Rehabilitation intervention for pwMS

INTERVENTIONS:
Behavioral: Vocational Rehabilitation intervention for pwMS — The VR intervention will cover three areas of intervention:
  * Rehabilitation Area: this intervention has the goal of managing the work performance from a rehabilitative point of view.
  * Reasonable accommodation area: this intervention has the goal of assessing the needs of reasonable accommodations, such has workspace modification, change in organization of the activities, management of work time, etc.., and propose it to the employer.
  * Educational and Formative Area: this area is responsible for the implementation of educational intervention for the employees and the employers about multiple sclerosis and its impact on work performance, the rights and obligations of the employer and employee about disability management on the workplace.

SUMMARY:
Multiple sclerosis (MS) is an autoimmune demyelinating disease of the central nervous system with both inflammatory and degenerative characteristics that affects approximately 136,000 people in Italy. The highest incidence of disease onset occurs between the ages of 20 and 40, which corresponds to the most productive period of a person's life. For this reason, one of the main social consequences of MS is the reduction or abandonment of work activity, which often begins in the early stages of the disease. Vocational Rehabilitation (VR) interventions, as reported in the literature, are used to manage and reduce work-related difficulties. The goal of VR is to enable individuals who experience difficulties in performing work activities to access, find, and maintain employment. This approach is characterized by its multi-professional and multidimensional nature, involving different types of interventions carried out by various professionals in diverse settings.

The overall aim of the project is to define a Vocational Rehabilitation (VR) protocol to reduce work-related challenges and promote job retention for workers with MS within the Italian healthcare and social context. The intervention will be organised into three different areas: rehabilitation, reasonable accommodation and education. Participants will receive any of the three interventions or a combination of these. The study will involve a multidisciplinary team of doctors (e.g. neurologist, physiatrist), psychologists, occupational therapists, physiotherapists, social workers, and labour law experts who will be involved according to the subject's specific needs.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed MS diagnosis
* Age ≥18 years
* Currently employed at the beginning of the study entry
* Have worked at least one day in the last 12 months
* MSQ-Job >=15
* Written informed consent

Exclusion Criteria:

* Presence of other pathologies impacting on work productivity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-01-15 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
Interception | Up to 6 months
  Number of eligible participants who has been invited to the VR intervention.
Acceptance | Up to 6 months
  Number of participants who accepts to be included in the VR intervention.
Adherence | Up to 6 months
  Number of participants who complete the VR intervention.
Lost to Follow-Up | Up to 6 months
  Number of dropouts from the VR intervention.
Canadian Occupational Performance Measure (COPM) | Baseline, up to 6 months
  The COPM employs a semi-structured interview that guides patients to define their concerns in three main areas: Self-care, Productivity - Paid or unpaid work, and Leisure. For the purposes of the study, only the "Paid or unpaid work" dimension will be assessed. Participants report two different scores regarding work activities' satisfaction and performance ranging from 1 to 10.
Client Satisfaction Questionnaire (CSQ) | Up to 6 months
  The Client Satisfaction Questionnaire collects data regarding satisfaction of participants on the VR intervention, using a 4 degree Likert scale ranging from one (not satisfied at all) to 4 (completly satisfied)
Global Perceived Effect (GPE) scale | Up to 6 months
  This is a patient reported rating scale commonly used in clinical and research settings. For the purposes of the study, it is used to assess the overall perception of effectiveness related to the global VR Intervention in terms of reduction of work difficulties. A scale likert ranging from 1 to 7, where 1 indicates the lowest perceived effectiveness of the intervention on work difficulties, and 7 the highest perceived effectiveness.
Barthel Index (BI) | Baseline, up to 6 months
  The scale measures the level of autonomy in the basic activity of daily living. It assesses ten different basic activities of daily living: using the toilet, bathing, bowel functions, dressing, eating, walking, climbing stairs and moving from bed to chair. By assessing each of these functions it is possible to calculate an autonomy index ranging from 0 (totally dependent) to 100 (totally independent)
Hospital Anxiety Depression scale (HADS) | Baseline, up to 6 months
  The scale assesses the presence of mood disorders. It is one of the most self-reported questionnaires widely used in the hospital and research context. Its aim is to screen for the presence of anxiety and depression. It consists of 14 items used to define two separate scores for anxiety and depression. For both scores there is a cut-off (8) useful for classifying the clinical condition of the patient as healthy or pathological.
Modified Fatigue (MFIS-21) | Baseline, up to 6 months
  The scale measures fatigue level. It consists of 21 items, which can be summed up to define 3 dimensions of fatigue: physical, cognitive and social. Subjects can respond to the items with a likert scale ranging from 0 (no fatigue) to 4 (highest level of fatigue)
Multiple Sclerosis Neuropsychological Questionnaire for patient (MSNQ-p) | Baseline, up to 6 months
  The questionnaire identifies possible participants at risk for cognitive impairment. This is a 15 self-reported outcome aimed to assess the presence of cognitive impairment in pwMS. Items covered different domain of cognitive functioning: processing speed, dual-task processing, attention, memory, executive function, and psychosocial comportment. The response scale ranges from 0 to 4, where 0 is "problem not encountered" and 4 "occurs very Frequently". A total maximum score of 60 is computed.
WHO Disability Assessment Schedule (WHODAS) | Baseline, up to 6 months
  The scale measures the impact of health conditions in daily life activities according to the Functioning, Disability and Health (ICF) framework. This questionnaire developed by the World Health Organization aimed to assess the impact of health status on client's level of functioning in six functional domains: cognition, mobility, self-care, getting along, life activities, participation. A score on a liker scale ranging from 1 to 5 indicates the impact of disability, with 1 indicating absence of impact and 5 the greatest possible impact. Each domain consists of five items. The score of each item are summed up to obtain a score for the individual functional domain. A total score is gained summing the total score of each functional domain.

CONTACTS AND LOCATIONS:
Overall Officials: Giampaolo Brichetto, PhD, Study Director — Fondazione Italiana Sclerosi Multipla
Locations (2):
- Italy (2):
  - IRCCS Fondazione Santa Lucia, Rome, Lazio
  - Servizio di Riabilitazione AISM Liguria, Italian Multiple Sclerosis Society, Genoa, Liguria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Vitturi BK, Rahmani A, Dini G, Montecucco A, Debarbieri N, Bandiera P, Ponzio M, Battaglia MA, Brichetto G, Inglese M, Persechino B, Durando P. Work Barriers and Job Adjustments of People with Multiple Sclerosis: A Systematic Review. J Occup Rehabil. 2023 Sep;33(3):450-462. doi: 10.1007/s10926-022-10084-1. Epub 2022 Nov 18. PMID 36399281
- [Background] Ponzio M, Pignattelli E, Verri A, Grange E, Persechino B, Vitturi BK, Bandiera P, Manacorda T, Inglese M, Durando P, Battaglia MA. Job Retention by People With Disabilities: A Qualitative Study of the Perspectives of People With Multiple Sclerosis. Med Lav. 2024 Jun 21;115(3):e2024018. doi: 10.23749/mdl.v115i3.15947. PMID 38922837
- [Background] Ponzio M, Podda J, Pignattelli E, Verri A, Persechino B, Vitturi BK, Bandiera P, Manacorda T, Inglese M, Durando P, Battaglia MA. Work Difficulties in People with Multiple Sclerosis. J Occup Rehabil. 2024 Sep;34(3):606-617. doi: 10.1007/s10926-023-10149-9. Epub 2023 Nov 3. PMID 37921967
- [Background] Sweetland J, Riazi A, Cano SJ, Playford ED. Vocational rehabilitation services for people with multiple sclerosis: what patients want from clinicians and employers. Mult Scler. 2007 Nov;13(9):1183-9. doi: 10.1177/1352458507078414. Epub 2007 Jul 10. PMID 17623726
- [Background] Escorpizo R, Reneman MF, Ekholm J, Fritz J, Krupa T, Marnetoft SU, Maroun CE, Guzman JR, Suzuki Y, Stucki G, Chan CC. A conceptual definition of vocational rehabilitation based on the ICF: building a shared global model. J Occup Rehabil. 2011 Jun;21(2):126-33. doi: 10.1007/s10926-011-9292-6. PMID 21328061